CLINICAL TRIAL: NCT05723094
Title: Effect of Low-Level Laser Therapy on Stability During Retention Phase After Orthodontic Treatment: A Randomized Controlled Trial.
Brief Title: Effect of Low-Level Laser Therapy on Stability During Retention Phase.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, WANG YANPEI, MD, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USM/JEPeM/22060411
Record Dates: First submitted 2023-01-15; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Orthodontic Retainers; Laser Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Retention Laser Group (LG) (Experimental): Before the orthodontic retention phase, the Ga-Al-As diode laser(Ilase, USA) was applied to the experimental group.
  Interventions: Radiation: Ga-Al-As diode laser (Ilase, USA)
- Retention Control Group (CG) (Placebo Comparator): Before the orthodontic retention phase, those who did not apply the Ga-Al-As diode laser (Ilase, USA) were the control group.
  Interventions: Other: placebo

INTERVENTIONS:
Radiation: Ga-Al-As diode laser (Ilase, USA) — The laser parameter used in previous study： Laser type：Ga-Al-As Wavelength：940 nm Emission type：Continuous Irradiation dosage/per tooth：75J/cm2 Application technique：Direct contact with the mucosa Exposure time per point：6 second Laser classification：3B Laser application time：Once in a month (4-week intervals) for the maxilla and mandibular incisors and canines Output：100Mw Diameter of the optical fiber：0.04 cm2
  Arms: Retention Laser Group (LG)
Other: placebo — Before the orthodontic retention phase, those who did not apply the Ga-Al-As diode laser (Ilase, USA) were the control group.
  Arms: Retention Control Group (CG)

SUMMARY:
The biggest problem in the orthodontic process is the pain and the long duration of treatment, which is also generally divided into 2 phases, namely the orthodontic tooth movement (OTM) and the retention phase. In recent decades, low-level-laser therapy has gained attention because it is non-invasive, inexpensive, relieves pain and has no significant adverse effects. Low-level-laser therapy (LLLT) has been proved to effectively induce and accelerate the remodeling process of alveolar bone by increasing the number of osteoblasts and osteoclasts. Therefore, LLLT is widely used in OTM to accelerate tooth displacement, but there are few studies and limited evidence on the stability whether it can strengthen and shorten the retention stage to avoid relapse. Thus, the purpose of this study is to investigate the stability after orthodontic treatment by observing the substantial influence of low-level-laser as during retention phase.

Research Question(s)

1. Does the low-level laser treatment can enhance stability and shorten retention time after orthodontic treatment or not will be demonstrated through 3 aspects：

1. The Incisor Irregularities Index between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention
2. The interarch dimension: intercanine width, intermolar width, interpremolar width, arch length between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention
3. The overjet and overbite between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention

Objective

General:

The goal of this study is to investigate the stability in retention phase after application of LLLT during leveling and alignment with fixed appliances.

Specific:

1. To compare the Incisor Irregularities Index between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention
2. To compare the interarch dimension: intercanine width, intermolar width, interpremolar width, arch length between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention To compare the overjet and overbite between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention

DETAILED DESCRIPTION:
This is a continuation study from the previous approved project entitle "The Effect of low level laser therapy on orthodontic tooth movement using conventional and self-ligating brackets in extractions cases: A randomised clinical trial and 3D evaluation via CBCT and digital dental model approaches" with ethical approval no ( USM/JEPeM/17070339). Previous studies used an in-vivo study, designed as randomised clinical trial for patients under treatment with fixed orthodontic brackets in Orthodontic Specialist Clinic at Hospital Universiti Sains Malaysia.

The current study was designed to observe the effect of laser irradiation (LLLT) during retention period at debond (0), 6 and 12 months of retention phases. The laser (LLLT dose) was applied only during active orthodontic treatment (levelling and alignment stage) in previous study. Patients will not receive any more doses of LLLT during retention phases at debond (0), 6 and 12 months.

All participants (control group and experimental group) from the previous studies will be included and enrolled in this current study after receiving the consent from patients. Among them, those who received LLLT in the previous study will be enrolled in the Retention Laser Group (LG) and those who did not receive LLLT will be in the Retention Control Group (CG) for the current study. The smaller the variation in tooth alignment between LG and CG, the better the retention stability.

In this current study, Little's Irregularity Index (LII), overjet, overbite, arch length, intermolar and intercuspid widths will be used as indicators for the stability assessment.

Study population The same participants from project entitle "The Effect of low level laser therapy on orthodontic tooth movement using conventional and self-ligating brackets in extractions cases: A randomised clinical trial and 3D evaluation via CBCT and digital dental model approaches" with ethical approval no (USM/JEPeM/17070339) treated at Specialist Orthodontic Clinic, Hospital Universiti Sains Malaysia will be recruited for this current study.

Sampling method and subject recruitment Patients who meet the inclusion and exclusion criteria and ready to debond will be invited to participate in this current trial. The orthodontist will have provided patients (≥18years) with verbal and written information about the study protocol in order to obtain the consent.

This study is a continuation of a previous research project as stated in the study design section where the sampling method used was simple random sampling. Previous research project was conducted in the Specialist Orthodontic Clinic, School of Dental Sciences, Hospital USM. A total of thirty-two patients were randomised using the online free randomisation software (http://www.randomization.com). The software automatically generated the randomisation plan where the number of patients were balanced in each group (1:1). Thus, the subjects were recruited in each group blindly following the randomisation plan. A total of sixteen patients were included in LLLT and non-LLLT groups, respectively. During the follow up, none of the patients were discontinued from each group. Therefore, a total of thirty-two patients will selected for the current study, those who received LLLT in the previous study will be enrolled in the Retention Laser Group (LG) and those who did not receive LLLT will be in the Retention Control Group (CG).

Operational definition

Study variables:

Independent variable is Retention laser group (LG), Retention control group (CG) and difference stages which is debond (0), 6 months and 12 months.

Dependent variable is LII index, arch lengh, intercanin length, intermolar width, overjet and overbite.

1. Little's Irregularity Index (LII, mm) A modification of Little's technique (Little, 1975), the sum of the distances between the anatomic contact points from the mesial of the left canine to the mesial of the right canine.
2. Arch length (left, mm) The distance between the incisal contact point of the central incisors to the mesial contact point of the left first permanent molar.
3. Arch length (right, mm) The distance between the incisal contact point of the central incisors to the mesial contact point of the right first permanent molar.
4. Arch length (total, mm) The sum of arch length (left) and arch length (right).
5. Intercanine width ICW, mm) The distance between the cusp tips of the permanent canines. In case of tooth abrasion, the midpoint of the plateau was used.
6. Intermolar width (IMW, mm) The distance between the mesiobuccal cusp tips of the left and right first permanent molars. In case of tooth abrasion, the midpoint of the plateau.
7. Overjet (OJ, mm) The distance of the most labial maxillary central incisor to the labial surface of the mandibular central incisor.
8. Overbite (OB, mm) The mean overlaps of the maxillary to the mandibular central incisors.

Data collection method and Research tools

1 Application of laser in the previous study. A Ga-Al-As diode laser (Ilase, USA) with a wavelength of 940 nm has been used in the previous study, operating in continuous wavelength (CW) mode. The fiber diameter of the laser beam is 0.04 cm2 (Figure 1.1). The tip of the optical fiber is kept in contact with the mucosa during irradiation. The laser was irradiated to five points on each dental site (Figure 1.2). The points are: two points in the mesial and distal apical regions, one point approximately in the middle of the cervical part of the incisor and canine (Figure 1.3). The conventional irradiation point is at the labial side of the maxillary and mandibular dental arches. The laser parameters that have been used in previous study are shown in (Table 1). The procedure was performed in an isolated room where the patient, the operator and the dental assistant wear the protective glasses. The energy density calculated on each tooth was calculated using the following equation: Energy density = laser output power x Sec / diameter in cm2.

Table 1: The laser parameter used in previous study:

Laser type: Ga-Al-As Wavelength: 940 nm Emission type : Continuous Irradiation dosage/per tooth: 75J/cm2 Application technique: Direct contact with the mucosa Exposure time per point: 6 second Laser classification: 3B Laser application time: Once in a month (4-week intervals) for the maxilla and mandibular incisors and canines Output: 100Mw Diameter of the optical fiber: 0.04 cm2

2. Specific operations for Retention Laser group (LG) and Retention Control group (CG) (1:1) After finishing the active orthodontic treatment and the patients ready for debonding (removal of braces), all participants from both groups LG and CG will be issues and wear the same type of retainer which is Vacuum formed retainer (VFR) during the retention phase. At debond (0), 6 and 12 months of retention phases, all patients will not receive any more doses of laser. All patients from both groups will be instructed to wear the retainer following the same regime as usual practice. Patients need to wear the VFR retainer for full time (24 hours daily) for 12 months of debonding and only remove the retainer during eating and brushing.

The VFR will be fabricated from copolyester material (Transparent Copyplast C, size 1.0x125mm) following the manufacture's instructions. It will be heated for 90 seconds then cool for 150 seconds with 0.5mm thickness after thermoformed. The retainer will be trimmed to provide 1-2 mm buccal and 3-4mm lingual extension past the gingival margins. All occlusal surfaces will be covered up to and included the most distal teeth.

3. Study model preparation and collections Alginate impression at debond (0) and after 6 and 12 months of retention after debonding will be obtained from participants. Then the dental cast will be fabricated using dental stone to produce a study model.

The series of the study models collected from patients according to intervention time will be scanned individually using scanner machine (Next Engine) to produce the 3D model for the measurements of the variables.

The Next Engine 3D laser scanner (Next Engine Inc, Canada) will be used to analyze the pre-and post-dental models for both groups for transverse dental changes and irregularities index.

The computer, scanner, and auto-drive are all included in the 3D scanner equipment. The gripper arm, platter pad, and platter shaft make up the auto drive. A platter pad may be used to carry the cast, and a gripper arm can be used to secure it. The platter pad screw can also be used to adjust the cast up, down, right, and left. The gripper arm is moved up and down by a screw. The scanner and the auto-drive are connected by a USB connection. Another USB cord connects the scanner to the computer. Scanning can be divided into three categories: scan family, placement, and divisions. To scan the cast from every angle, select the 360-degree scan option from the panel. The next-generation 3D laser scanner can detect an object's length, width, and depth by triangulating distances between the reflecting aser beam and the scanned cast surface.

The following engine, the 3D laser scanner, uses a Class II laser gamma of 685 nm at 25 mW, with a beam-spread angle (2 Theta) of 21 horizontally and 0.1 vertically, an object-to-scanner distance of 0.3 m, a field of view of 70 mm, and a scanning time of 30 seconds. For its 3D data, the scanner uses a one-half-inch frame transfer charged coupled device (CCD) with 380,000 pixels, as well as a color CCD with a similar specification. The output data from the scanner is 200 x 200 x 256 for 3D and 400 x 400 for color data. The device weighs one kilogram in total.

All scanned data coordinates (in x, y, and z) are imported in DXF format into ScanStudio HD software to be measured. Spatial linear measurements are taken using a digital caliper (computer mouse) that is accurate to 0.5 mm, and the average value is used.

Blinding

The clinician and researcher will be blinding because both groups use the same type of retainers and the impression will be taken at the same time frame. Furthermore, no more laser dose will be given during the retention period.

Questionnaires A set of questionnaires will be distributed to the participants at the end of the final data collections at 12 months of retention phase to assess the patients' compliances. The questionnaires used for this study was adapted from the questionnaire used by Ab Rahman et al with permission. The questionnaires will be available in both languages; English and Malay and the version will be given according to participant preference in term of language.

Community sensitivities and benefits If the result from this current study shows the LG group proven to have a better stability during the retention phase, some suggestions can be provided to the orthodontists/clinician such as to use the LLLT during the active orthodontic treatment not only to shorten the treatment duration and reduce the pain during active treatment but the laser also can obtained more stability after debonding. Another advantages, the duration/ regime to wear the retainer can be shorten to avoid burden of the patients in wearing the retainer.

Data analysis Descriptive statistics will be calculated for each measurement (mean, median, standard deviation, and Inter-Quartile Range). The amount of relapse will be described by comparing the measurements at the time of debonding (T1), after 6 months (T2), and after 12 months (T3) of wear of the retainer. Data were analysed using Statistical Package for the Social Sciences (SPSS) version 26. One-way repeated measure ANOVA will be used to compare the Incisor Irregularities Index between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention (Objective 1). Two-way repeated measure ANOVA will be used to compare the interarch dimension: intercanine width, intermolar width, interpremolar width, arch length, overjet and overbite between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention (Objective 2 and Objective 3). The level of significance for the statistical analysis is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patient treated with laser and non-laser application during orthodontic treatment as in previous study
* 2.The patient presents with mild to moderate crowding malocclusion with extraction of all 1st premolars and using conventional brackets
* 3.The treatment of fixed appliances involving both arches
* 4. Patients wearing vacuum formed retainers.
* 5. Patients are compliance towards retainer wear with no history of retainer lost
* 6. All permanent teeth erupted except for third molars.

Exclusion Criteria:

* 1.Age less than 18 years old
* 2.Active caries and Periodontal disease
* 3.Use any long-term use of analgesics or drugs that affect the function of the central nervous system.
* 4. Non-compliance patients in term of wearing retainers

Withdrawal criteria:

* 1.Any patient who would like to withdraw from the experiment can do without their treatment being compromised.
* 2.Patients who do not comply with the retainer requirements during the retention phase will be considered an automatic withdrawal from the research and their data will not be accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-12-18 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Incisor Irregularities Index | 12 months
  To compare the changes in the Incisor Irregularities Index between the laser and control group after the application of LLLT at debond (0), 6, and 12 months of retention.
The interarch dimension: intercanine width, intermolar width, interpremolar width, arch length | 12 months
  To compare the changes in the interarch dimension: intercanine width, intermolar width, interpremolar width, arch length between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention
Overjet and overbite | 12 months
  To compare the changes in the overjet and overbite between laser and control group after application of LLLT at debond (0), 6 and 12 months of retention

CONTACTS AND LOCATIONS:
Overall Officials: Norma Binti Ab Rahman, MASTER, Study Director — SCHOOL OF DENTAL SCIENCES
Locations (1):
- Wang Yanpei, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ab Rahman N, Wey MC, Othman SA. Mandibular arch orthodontic treatment stability using passive self-ligating and conventional systems in adults: A randomized controlled trial. Korean J Orthod. 2017 Jan;47(1):11-20. doi: 10.4041/kjod.2017.47.1.11. Epub 2016 Dec 19. PMID 28127535
- [Background] Abi-Ramia LB, Stuani AS, Stuani AS, Stuani MB, Mendes Ade M. Effects of low-level laser therapy and orthodontic tooth movement on dental pulps in rats. Angle Orthod. 2010 Jan;80(1):116-22. doi: 10.2319/120808-619.1. PMID 19852650
- [Background] Akin E, Gurton AU, Olmez H. Effects of nitric oxide in orthodontic tooth movement in rats. Am J Orthod Dentofacial Orthop. 2004 Nov;126(5):608-14. doi: 10.1016/S0889540604004494. PMID 15520694
- [Background] Bjordal JM, Lopes-Martins RA, Iversen VV. A randomised, placebo controlled trial of low level laser therapy for activated Achilles tendinitis with microdialysis measurement of peritendinous prostaglandin E2 concentrations. Br J Sports Med. 2006 Jan;40(1):76-80; discussion 76-80. doi: 10.1136/bjsm.2005.020842. PMID 16371497
- [Background] Boldrini C, de Almeida JM, Fernandes LA, Ribeiro FS, Garcia VG, Theodoro LH, Pontes AE. Biomechanical effect of one session of low-level laser on the bone-titanium implant interface. Lasers Med Sci. 2013 Jan;28(1):349-52. doi: 10.1007/s10103-012-1167-3. Epub 2012 Jul 24. PMID 22825319
- [Background] Burke SP, Silveira AM, Goldsmith LJ, Yancey JM, Van Stewart A, Scarfe WC. A meta-analysis of mandibular intercanine width in treatment and postretention. Angle Orthod. 1998 Feb;68(1):53-60. doi: 10.1043/0003-3219(1998)0682.3.CO;2. PMID 9503135
- [Background] Burstone CR. Deep overbite correction by intrusion. Am J Orthod. 1977 Jul;72(1):1-22. doi: 10.1016/0002-9416(77)90121-x. PMID 267433
- [Background] Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR. The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. 2012 Feb;40(2):516-33. doi: 10.1007/s10439-011-0454-7. Epub 2011 Nov 2. PMID 22045511
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Doshi-Mehta G, Bhad-Patil WA. Efficacy of low-intensity laser therapy in reducing treatment time and orthodontic pain: a clinical investigation. Am J Orthod Dentofacial Orthop. 2012 Mar;141(3):289-297. doi: 10.1016/j.ajodo.2011.09.009. PMID 22381489
- [Background] Edman Tynelius G, Bondemark L, Lilja-Karlander E. A randomized controlled trial of three orthodontic retention methods in Class I four premolar extraction cases -- stability after 2 years in retention. Orthod Craniofac Res. 2013 May;16(2):105-15. doi: 10.1111/ocr.12011. Epub 2013 Jan 3. PMID 23324112
- [Background] Franzen TJ, Monjo M, Rubert M, Vandevska-Radunovic V. Expression of bone markers and micro-CT analysis of alveolar bone during orthodontic relapse. Orthod Craniofac Res. 2014 Nov;17(4):249-58. doi: 10.1111/ocr.12050. Epub 2014 Jun 15. PMID 24931826
- [Background] Franzen TJ, Brudvik P, Vandevska-Radunovic V. Periodontal tissue reaction during orthodontic relapse in rat molars. Eur J Orthod. 2013 Apr;35(2):152-9. doi: 10.1093/ejo/cjr127. Epub 2011 Oct 24. PMID 22023883
- [Background] Fujiyama K, Deguchi T, Murakami T, Fujii A, Kushima K, Takano-Yamamoto T. Clinical effect of CO(2) laser in reducing pain in orthodontics. Angle Orthod. 2008 Mar;78(2):299-303. doi: 10.2319/033007-153.1. PMID 18251609
- [Background] Gardner RB. A comparison of four methods of predicting arch length. Am J Orthod. 1979 Apr;75(4):387-98. doi: 10.1016/0002-9416(79)90160-x. PMID 285614
- [Background] Goldie RS, King GJ. Root resorption and tooth movement in orthodontically treated, calcium-deficient, and lactating rats. Am J Orthod. 1984 May;85(5):424-30. doi: 10.1016/0002-9416(84)90163-5. PMID 6586081
- [Background] Han G, Chen Y, Hou J, Liu C, Chen C, Zhuang J, Meng W. Effects of simvastatin on relapse and remodeling of periodontal tissues after tooth movement in rats. Am J Orthod Dentofacial Orthop. 2010 Nov;138(5):550.e1-7; discussion 550-1. doi: 10.1016/j.ajodo.2010.04.026. PMID 21055594
- [Background] Haruyama N, Igarashi K, Saeki S, Otsuka-Isoya M, Shinoda H, Mitani H. Estrous-cycle-dependent variation in orthodontic tooth movement. J Dent Res. 2002 Jun;81(6):406-10. doi: 10.1177/154405910208100610. PMID 12097433
- [Background] Hashimoto F, Kobayashi Y, Mataki S, Kobayashi K, Kato Y, Sakai H. Administration of osteocalcin accelerates orthodontic tooth movement induced by a closed coil spring in rats. Eur J Orthod. 2001 Oct;23(5):535-45. doi: 10.1093/ejo/23.5.535. PMID 11668873
- [Background] Hassan AH, Al-Hubail A, Al-Fraidi AA. Bone inductive proteins to enhance postorthodontic stability. Angle Orthod. 2010 Nov;80(6):1051-60. doi: 10.2319/112409-665.1. PMID 20677954
- [Background] Hirate Y, Yamaguchi M, Kasai K. Effects of relaxin on relapse and periodontal tissue remodeling after experimental tooth movement in rats. Connect Tissue Res. 2012;53(3):207-19. doi: 10.3109/03008207.2011.628060. Epub 2011 Dec 5. PMID 22141456
- [Background] Hudson JB, Hatch N, Hayami T, Shin JM, Stolina M, Kostenuik PJ, Kapila S. Local delivery of recombinant osteoprotegerin enhances postorthodontic tooth stability. Calcif Tissue Int. 2012 Apr;90(4):330-42. doi: 10.1007/s00223-012-9579-4. Epub 2012 Mar 1. PMID 22382900
- [Background] Sikorska A, Cudzilo D, Matthews-Kozanecka M, Turska-Malinska R. Impact of incorrect oral habits on mastication anomalies in children and adolescents - literature review and own observations. Dev Period Med. 2016;20(4):325-327. PMID 28216487
- [Background] Jones M, Chan C. The pain and discomfort experienced during orthodontic treatment: a randomized controlled clinical trial of two initial aligning arch wires. Am J Orthod Dentofacial Orthop. 1992 Oct;102(4):373-81. doi: 10.1016/0889-5406(92)70054-e. PMID 1456222
- [Background] Kale S, Kocadereli I, Atilla P, Asan E. Comparison of the effects of 1,25 dihydroxycholecalciferol and prostaglandin E2 on orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2004 May;125(5):607-14. doi: 10.1016/j.ajodo.2003.06.002. PMID 15127030
- [Background] Kanzaki H, Chiba M, Shimizu Y, Mitani H. Periodontal ligament cells under mechanical stress induce osteoclastogenesis by receptor activator of nuclear factor kappaB ligand up-regulation via prostaglandin E2 synthesis. J Bone Miner Res. 2002 Feb;17(2):210-20. doi: 10.1359/jbmr.2002.17.2.210. PMID 11811551
- [Background] Kawasaki K, Shimizu N. Effects of low-energy laser irradiation on bone remodeling during experimental tooth movement in rats. Lasers Surg Med. 2000;26(3):282-91. doi: 10.1002/(sici)1096-9101(2000)26:33.0.co;2-x. PMID 10738291
- [Background] Kim SJ, Kang YG, Park JH, Kim EC, Park YG. Effects of low-intensity laser therapy on periodontal tissue remodeling during relapse and retention of orthodontically moved teeth. Lasers Med Sci. 2013 Jan;28(1):325-33. doi: 10.1007/s10103-012-1146-8. Epub 2012 Jul 20. PMID 22814894
- [Background] Kim TW, Yoshida Y, Yokoya K, Sasaki T. An ultrastructural study of the effects of bisphosphonate administration on osteoclastic bone resorption during relapse of experimentally moved rat molars. Am J Orthod Dentofacial Orthop. 1999 Jun;115(6):645-53. doi: 10.1016/s0889-5406(99)70290-8. PMID 10358247
- [Background] King GJ, Thiems S. Chemical mediation of bone resorption induced by tooth movement in the rat. Arch Oral Biol. 1979;24(10-11):811-5. doi: 10.1016/0003-9969(79)90043-8. No abstract available. PMID 295604
- [Background] Kuijpers-Jagtman AM. [Repair and revision 8. Relapse of lower incisors: retreatment?]. Ned Tijdschr Tandheelkd. 2002 Feb;109(2):42-6. Dutch. PMID 11933564
- [Background] Lavine L, Lustrin I, Rinaldi R, Shamos M. Clinical and ultrastructural investigations of electrical enhancement of bone healing. Ann N Y Acad Sci. 1974;238:552-63. doi: 10.1111/j.1749-6632.1974.tb26821.x. No abstract available. PMID 4548337
- [Background] Limpanichkul W, Godfrey K, Srisuk N, Rattanayatikul C. Effects of low-level laser therapy on the rate of orthodontic tooth movement. Orthod Craniofac Res. 2006 Feb;9(1):38-43. doi: 10.1111/j.1601-6343.2006.00338.x. PMID 16420273
- [Background] Little RM. The irregularity index: a quantitative score of mandibular anterior alignment. Am J Orthod. 1975 Nov;68(5):554-63. doi: 10.1016/0002-9416(75)90086-x. PMID 1059332
- [Background] Luppanapornlarp S, Kajii TS, Surarit R, Iida J. Interleukin-1beta levels, pain intensity, and tooth movement using two different magnitudes of continuous orthodontic force. Eur J Orthod. 2010 Oct;32(5):596-601. doi: 10.1093/ejo/cjp158. Epub 2010 Jun 9. PMID 20534713
- [Background] Kreisler M, Christoffers AB, Willershausen B, d'Hoedt B. Effect of low-level GaAlAs laser irradiation on the proliferation rate of human periodontal ligament fibroblasts: an in vitro study. J Clin Periodontol. 2003 Apr;30(4):353-8. doi: 10.1034/j.1600-051x.2003.00001.x. PMID 12694435
- [Background] McNamara DC. Pathophysiology of occlusal balance. Aust Dent J. 1976 Jun;21(3):247-51. doi: 10.1111/j.1834-7819.1976.tb05758.x. PMID 1068685
- [Background] Mohammed AH, Tatakis DN, Dziak R. Leukotrienes in orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 1989 Mar;95(3):231-7. doi: 10.1016/0889-5406(89)90053-x. PMID 2538053
- [Background] Nanda RS, Nanda SK. Considerations of dentofacial growth in long-term retention and stability: is active retention needed? Am J Orthod Dentofacial Orthop. 1992 Apr;101(4):297-302. doi: 10.1016/S0889-5406(05)80321-X. PMID 1558058
- [Background] Ngan P, Kess B, Wilson S. Perception of discomfort by patients undergoing orthodontic treatment. Am J Orthod Dentofacial Orthop. 1989 Jul;96(1):47-53. doi: 10.1016/0889-5406(89)90228-x. PMID 2750720
- [Background] Nguyen QV, Bezemer PD, Habets L, Prahl-Andersen B. A systematic review of the relationship between overjet size and traumatic dental injuries. Eur J Orthod. 1999 Oct;21(5):503-15. doi: 10.1093/ejo/21.5.503. PMID 10565091
- [Background] Ong CK, Walsh LJ, Harbrow D, Taverne AA, Symons AL. Orthodontic tooth movement in the prednisolone-treated rat. Angle Orthod. 2000 Apr;70(2):118-25. doi: 10.1043/0003-3219(2000)0702.0.CO;2. PMID 10832999
- [Background] Qamruddin I, Alam MK, Mahroof V, Fida M, Khamis MF, Husein A. Effects of low-level laser irradiation on the rate of orthodontic tooth movement and associated pain with self-ligating brackets. Am J Orthod Dentofacial Orthop. 2017 Nov;152(5):622-630. doi: 10.1016/j.ajodo.2017.03.023. PMID 29103440
- [Background] Coombe AR, Ho CT, Darendeliler MA, Hunter N, Philips JR, Chapple CC, Yum LW. The effects of low level laser irradiation on osteoblastic cells. Clin Orthod Res. 2001 Feb;4(1):3-14. doi: 10.1034/j.1600-0544.2001.040102.x. PMID 11553080
- [Background] Ren Y, Maltha JC, Van 't Hof MA, Kuijpers-Jagtman AM. Optimum force magnitude for orthodontic tooth movement: a mathematic model. Am J Orthod Dentofacial Orthop. 2004 Jan;125(1):71-7. doi: 10.1016/j.ajodo.2003.02.005. PMID 14718882
- [Background] Saito S, Shimizu N. Stimulatory effects of low-power laser irradiation on bone regeneration in midpalatal suture during expansion in the rat. Am J Orthod Dentofacial Orthop. 1997 May;111(5):525-32. doi: 10.1016/s0889-5406(97)70152-5. PMID 9155812
- [Background] Sonesson M, De Geer E, Subraian J, Petren S. Efficacy of low-level laser therapy in accelerating tooth movement, preventing relapse and managing acute pain during orthodontic treatment in humans: a systematic review. BMC Oral Health. 2016 Jul 7;17(1):11. doi: 10.1186/s12903-016-0242-8. PMID 27431504
- [Background] Staley RN, Stuntz WR, Peterson LC. A comparison of arch widths in adults with normal occlusion and adults with class II, Division 1 malocclusion. Am J Orthod. 1985 Aug;88(2):163-9. doi: 10.1016/0002-9416(85)90241-6. PMID 3861102
- [Background] Torri S, Weber JB. Influence of low-level laser therapy on the rate of orthodontic movement: a literature review. Photomed Laser Surg. 2013 Sep;31(9):411-21. doi: 10.1089/pho.2013.3497. Epub 2013 Jul 24. PMID 23883115
- [Background] Tortamano A, Lenzi DC, Haddad AC, Bottino MC, Dominguez GC, Vigorito JW. Low-level laser therapy for pain caused by placement of the first orthodontic archwire: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2009 Nov;136(5):662-7. doi: 10.1016/j.ajodo.2008.06.028. PMID 19892282
- [Background] Tyrovola JB, Spyropoulos MN. Effects of drugs and systemic factors on orthodontic treatment. Quintessence Int. 2001 May;32(5):365-71. PMID 11444068
- [Background] Wakabayashi H, Hamba M, Matsumoto K, Tachibana H. Effect of irradiation by semiconductor laser on responses evoked in trigeminal caudal neurons by tooth pulp stimulation. Lasers Surg Med. 1993;13(6):605-10. doi: 10.1002/lsm.1900130603. PMID 8295468
- [Background] Wu S, Chen Y, Zhang J, Chen W, Shao S, Shen H, Zhu L, Ye P, Svensson P, Wang K. Effect of low-level laser therapy on tooth-related pain and somatosensory function evoked by orthodontic treatment. Int J Oral Sci. 2018 Jul 2;10(3):22. doi: 10.1038/s41368-018-0023-0. PMID 29967411
- [Background] Xie H, Bendre SC, Burke AP, Gregory KW, Furnary AP. Laser-assisted vascular end to end anastomosis of elastin heterograft to carotid artery with an albumin stent: a preliminary in vivo study. Lasers Surg Med. 2004;35(3):201-5. doi: 10.1002/lsm.20092. PMID 15389735
- [Background] Yoshida T, Yamaguchi M, Utsunomiya T, Kato M, Arai Y, Kaneda T, Yamamoto H, Kasai K. Low-energy laser irradiation accelerates the velocity of tooth movement via stimulation of the alveolar bone remodeling. Orthod Craniofac Res. 2009 Nov;12(4):289-98. doi: 10.1111/j.1601-6343.2009.01464.x. PMID 19840281
- [Background] Yoshida Y, Sasaki T, Yokoya K, Hiraide T, Shibasaki Y. Cellular roles in relapse processes of experimentally-moved rat molars. J Electron Microsc (Tokyo). 1999;48(2):147-57. doi: 10.1093/oxfordjournals.jmicro.a023661. PMID 10356787
- [Background] Zengo AN, Pawluk RJ, Bassett CA. Stress-induced bioelectric potentials in the dentoalveolar complex. Am J Orthod. 1973 Jul;64(1):17-27. doi: 10.1016/0002-9416(73)90277-7. No abstract available. PMID 4515022
- [Background] Zhao N, Lin J, Kanzaki H, Ni J, Chen Z, Liang W, Liu Y. Local osteoprotegerin gene transfer inhibits relapse of orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2012 Jan;141(1):30-40. doi: 10.1016/j.ajodo.2011.06.035. PMID 22196183